CLINICAL TRIAL: NCT03875833
Title: Prospective Analysis of Effect of Collagen Wrap Conduit on Radial and Ulnar Nerve Function Following Radial/Ulnar Forearm Free Flap Harvest
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, James C Melville, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-DB-18-0760
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Neoplasms; Dysesthesia
MeSH Terms: conditions — Head and Neck Neoplasms; Paresthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Collagen Nerve Wrap Conduit (Experimental)
  Interventions: Device: Collagen Nerve Wrap Conduit
- Control (No Intervention)

INTERVENTIONS:
Device: Collagen Nerve Wrap Conduit — The collagen nerve wrap conduit will be placed on all exposed radial and ulnar nerves at the time of free flap harvest.
  Arms: Collagen Nerve Wrap Conduit

SUMMARY:
The purpose of this study is to determine whether collagen nerve conduits placed on exposed radial and ulnar nerves during radial and ulnar forearm free flap harvests will reduce the occurrence and degree of sensory nerve deficit.

ELIGIBILITY:
Inclusion Criteria:

* patients present with a complex defect after tumor resection
* all these cases done with the departments of Oral and Maxillofacial Surgery and Otolaryngology at the University of Texas in multiple locations that include, Memorial Hermann Hospital, Ben Taub General Hospital, Lyndon B. Johnson General Hospital and The Methodist hospital.
* patients that have been diagnosed with head and neck tumors and who will undergo a composite resection and reconstruction with radial or ulnar free vascularized flap.

Exclusion Criteria:

* pre-existing nerve deficits
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with normal sensory recovery at the site of forearm free flap as assessed by subjective patient questionnaire regarding upper extremity sensation and function | baseline
Number of participants with normal sensory recovery at the site of forearm free flap as assessed by subjective patient questionnaire regarding upper extremity sensation and function | 3 months
Number of participants with normal sensory recovery at the site of forearm free flap as assessed by subjective patient questionnaire regarding upper extremity sensation and function | 6 months
Number of participants with normal sensory recovery at the site of forearm free flap as assessed by subjective patient questionnaire regarding upper extremity sensation and function | 12 months
Number of participants with normal sensory recovery at the site of forearm free flap as assessed by objective clinical findings | baseline
  Participants will be evaluated clinically using pinprick, light touch, and two-point discrimination tests. An overall score will be reported.
Number of participants with normal sensory recovery at the site of forearm free flap as assessed by objective clinical findings | 3 months
  Participants will be evaluated clinically using pinprick, light touch, and two-point discrimination tests. An overall score will be reported.
Number of participants with normal sensory recovery at the site of forearm free flap as assessed by objective clinical findings | 6 months
  Participants will be evaluated clinically using pinprick, light touch, and two-point discrimination tests. An overall score will be reported.
Number of participants with normal sensory recovery at the site of forearm free flap as assessed by objective clinical findings | 12 months
  Participants will be evaluated clinically using pinprick, light touch, and two-point discrimination tests. An overall score will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: James C Melville, DDS, Principal Investigator — The University of Texas Health Science Center, Houston

IPD SHARING:
Plan to Share IPD: No